CLINICAL TRIAL: NCT03375112
Title: Pain Control After Total Hip Arthroplasty: A Randomized Trial Determining Efficacy of Fascia Iliaca Compartment Blocks in the Immediate Post-Operative Period
Brief Title: Fascia Iliaca Blocks for Pain Control After Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Michael Charters, MD, Orthopac Surgeon, Department of Joint Replacement and Reconstruction, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: FICB01
Record Dates: First submitted 2017-03-22; First posted 2017-12-15 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Arthritis of Hip
Keywords: Total Hip Arthroplasty; Fascia Iliaca; Nerve Block; Pain Control
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be randomized to receive fascia iliaca blocks post-operatively or to receive a touch with a blunt needle and a bandaid post-operatively by the regional anesthesia team. Neither the patient nor the investigators will have knowledge of which group the patients belong to until the completion of the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fascia Iliaca Compartment Block (Experimental): A Fascia Iliaca Compartment Block will be administered in the block room.
  Interventions: Procedure: Fascia iliaca compartment block; Drug: Bupivacaine
- Control (Placebo Comparator): The patients will be brought back to the block room, prepped, and a blunt needle will be touched to the skin. A band aid will be applied over the site.
  Interventions: Drug: Placebo

INTERVENTIONS:
Procedure: Fascia iliaca compartment block — The patient will be brought to the block room within 30 minutes of arriving in recovery. An injection of local anesthetic into the fascia iliaca compartment using ultrasound guidance will be administered. The patient will then be transported back to recovery.
  Arms: Fascia Iliaca Compartment Block
Drug: Placebo — The patient will be brought to the block room within 30 minutes of arriving in recovery. An ultrasound probe will be placed to the skin and a blunt needle will be touched to the patient's skin in the area that a fascia iliaca compartment block would be performed. The patient will then be transported back to recovery.
  Arms: Control
Drug: Bupivacaine — A one time dose of 40 milliliters of 0.5% bupivacaine will be injected into the fascia iliaca compartment
  Arms: Fascia Iliaca Compartment Block

SUMMARY:
The fascia iliaca compartment block (FICB) is a regional block that anesthetizes the femoral, obturator, and lateral femoral cutaneous nerves around the hip. The purpose of this study is to determine whether FICB can reduce postoperative pain and increase progress with physical therapy after total hip arthroplasty (THA). This randomized, double-blind, clinical trial will randomize patients to receive either a FICB or placebo after THA. The primary outcomes will be pain scores reported by the patient post-operatively.

DETAILED DESCRIPTION:
The FICB is a regional block that anesthetizes the femoral, obturator, and lateral femoral cutaneous nerves around the hip joint. There have been numerous study assessing it's ability to control pain in the pre and post operative period in patients with hip fractures. However, there is a limited amount of literature on its efficacy after total hip arthroplasty, and no data when a posterior surgical approach to the hip was utilized. Because regional blocks have been shown to decrease pain post operatively after total knee arthroplasty, we hypothesize that the FICB will decrease pain and narcotic use in patients after total hip arthroplasty. This study will aim to recruit 120 patients that will be randomized to receive a FICB or placebo in the recovery room within 30 minutes of leaving the OR. Once the intervention is complete we will collect data on the patients' pain levels, morphine equivalents of narcotic that they used, and how well they worked with physical therapy during their inpatient stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Scheduled for total hip arthroplasty at Henry Ford Hospital
* Epidural anesthesia during surgery

Exclusion Criteria:

* Pregnancy
* Known intolerance to local anesthetic or narcotics
* Revision hip surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Charters, MD, Principal Investigator — Henry Ford Hospital
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bober K, Kadado A, Charters M, Ayoola A, North T. Pain Control After Total Hip Arthroplasty: A Randomized Controlled Trial Determining Efficacy of Fascia Iliaca Compartment Blocks in the Immediate Postoperative Period. J Arthroplasty. 2020 Jun;35(6S):S241-S245. doi: 10.1016/j.arth.2020.02.020. Epub 2020 Feb 14. PMID 32222267

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fascia Iliaca Compartment Block | Control
Started | 62 | 60
Completed | 59 | 60
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fascia Iliaca Compartment Block | Control | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.9 (12.8) | 63.6 (10.3) | 63.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 28 | 24 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary Osteoarthritis [Count of Participants; unit: Participants] | 57 | 59 | 116
Smoking [Count of Participants; unit: Participants] | 2 | 3 | 5
Prior Opioids use [Count of Participants; unit: Participants] | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Averaged Pain Score
Description: Analog pains scale 0-10. A pain score of 10 represents maximum pain and a pain score of 0 represents no pain.
Time Frame: Pain scores were at 30 minute intervals for the first hour post-operative, hourly for the next 4 hours, 2 hour intervals for the next 12 hours, then at 4 hour intervals until the 48 hour post-operative or discharge. The mean of these scores is reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Fascia Iliaca Compartment Block | Control
Number analyzed (Participants) | 59 | 60
score on a scale | 3.75 [3.5 to 5.8] | 4.11 [1.9 to 5]

2. Primary Outcome: Morphine Equivalents Consumed
Description: Total morphine equivalents (consumed at 4-hour time intervals) received in postoperative inpatient stay.
Time Frame: Postoperative inpatient stay, which averages approximately two days.
Measure: Mean (Standard Deviation); unit: morphine milliequivalents
Arm/Group | Fascia Iliaca Compartment Block | Control
Number analyzed (Participants) | 59 | 60
morphine milliequivalents | 75.3 (43.4) | 86.0 (55.6)

3. Secondary Outcome: Walking Distance
Description: The distance the patient is able to walk with physical therapy during their first session
Time Frame: Post operative day one
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Fascia Iliaca Compartment Block | Control
Number analyzed (Participants) | 59 | 60
Feet | 67.1 (59.1) | 68.3 (54.0)

4. Secondary Outcome: Time to Up-and-go
Description: Time to up and go test performed on the first postoperative day. This test is administered by having the patient sit in a chair. When the patient is instructed to start, the stand from the chair, walk to a marker ten feet away from the chair, turn around, return to the chair, and sit back down. The time is measured as the time from when the start command is given to when they are returned to a seated position.
Time Frame: Post operative day one
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Fascia Iliaca Compartment Block | Control
Number analyzed (Participants) | 59 | 60
Seconds | 63.7 (62.8) | 66.3 (63.9)

5. Secondary Outcome: Time to Discharge Readiness
Description: Time in hours since surgery to when the patient's pain is controlled on oral medications, has cleared physical and occupational therapy, and has no medical issues that require inpatient treatment.
Time Frame: Every 6 hours after surgery until completion of inpatient stay, an average of two days days after surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fascia Iliaca Compartment Block | Control
Number analyzed (Participants) | 59 | 60
hours | 35.1 (12.8) | 35.2 (11.8)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the initial inpatient recovery period (up to postoperative day 2), and during the routine follow-up clinical visits (at two weeks and six weeks).
Arm/Group | Fascia Iliaca Compartment Block | Control
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 0/59 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT03375112/Prot_SAP_002.pdf